CLINICAL TRIAL: NCT04562636
Title: Evaluating a Messaging Campaign in the United States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-2552; 14380 (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Heart Diseases; Cancer
Keywords: Red meat; Processed meat; Sustainability; Meat reduction
MeSH Terms: conditions — Obesity; Heart Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Environment-focused Meatless Monday messages (Experimental): Four environmental messages from the Meatless Monday campaign.
  Interventions: Other: Environmental message
- Health-focused Meatless Monday messages (Experimental): Four health messages from the Meatless Monday campaign.
  Interventions: Other: Health message
- Neutral Message (Other): Four neutral messages about checking one's credit score.
  Interventions: Other: Neutral Message

INTERVENTIONS:
Other: Environmental message — Participants will be randomized to view a set of four messages about the environmental harms of meat production from the Meatless Monday campaign.
  Arms: Environment-focused Meatless Monday messages
Other: Health message — Participants will be randomized to view a set of four messages about the health harms of meat consumption from the Meatless Monday campaign.
  Arms: Health-focused Meatless Monday messages
Other: Neutral Message — Participants will be randomized to view a set of four messages about checking their credit score.
  Arms: Neutral Message

SUMMARY:
Purpose: To evaluate reactions to and opinions of a messaging campaign.

Participants: Participants will be recruited through Prime Panels and will be US-based adults (18 years old and older) who consumed red meat in the past 30 days.

Procedures (methods): After completing a screening question about meat consumption, participants will review a consent form. If they select to participate in the study, participants will be randomly assigned to view control messages, red meat-related environment messages, or red meat-related health messages. They will be asked a series of questions about these messages.

Participants will also be asked about grocery shopping preferences and standard demographics questions.

DETAILED DESCRIPTION:
Excess consumption of red and processed meat is a growing problem, especially in the United States where meat is consumed more than three times the global average. Epidemiological evidence for the association between excess meat intake and negative health outcomes (such as cancer, cardiovascular disease, and type 2 diabetes) as well as negative environmental impacts (such as pollution, overuse of resources, and carbon emissions) indicates that reducing meat consumption should be particularly pertinent to researchers and other public health professionals.

The potential of using widespread communication campaigns, such as Meatless Monday, to reduce meat consumption by educating individuals on the associated health and environmental risks appears to be promising. However, the current literature is missing information regarding what types of messages are most effective (e.g. negative environmental messages vs. negative health messages). To address this knowledge gap, our study will collect quantitative data in measurable outcomes to understand effectiveness and comprehension of environmental messages and health messages to reduce meat consumption.

Setting: This is an online study using Qualtrics, so this research does not involve talking to human participants.

Recruitment: Participants will be recruited through Prime Panels, a survey research firm through which participants voluntarily sign up to participate in research studies.

Informed Consent: Participants will read a written consent document that includes information about the study's purpose, expectations, and possible risks and benefits. Participants will acknowledge that they have read and agreed to the terms by clicking forward.

Randomization: Participants will be randomly assigned to one of three groups: 1) control (about checking their credit score), 2) environment-focused Meatless Monday messages, or 3) health-focused Meatless Monday messages.

Assessment: Using an online platform (Qualtrics), participants will answer a screening question about red meat consumption. If they are eligible (consumption of red meat 1 time per week or more), they will proceed to the main study after reading and agreeing to the written consent form. Participants will then answer two questions about their belief in climate change. Participants will then view four messages in their ascribed conditions. After viewing all 4 messages, participants will answer a series of questions about the messages they viewed. Then, participants will answer a series of demographic questions. Participants will also answer questions about grocery shopping preferences.

Detailed description of the trial arms: This study is a three-armed between subjects' design. Participants will be randomized to view a set of four messages either about the environmental harms of meat production (intervention), the health harms of meat consumption (intervention), or about checking their credit score (control). The environmental and health harms messages were obtained from existing publicly available messages from the Meatless Monday campaign.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Be able to read and speak English
* Be able to take a computer survey in English
* Currently reside in the United States
* Consumed red meat in the past 30 days

Exclusion Criteria:

* Non red-meat eater

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1244 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Perceived Message Effectiveness (PME) | ~10 minute computer survey immediately after seeing messages
  Perceived effectiveness of the messages will be measured during the message using 4 items adapted from Baig et al. (2018): concern, unpleasantness, and discouragement. The averaged responses on the 4 items will be used to create a PME score. All 4 items are measured using a a 1 to 5 likert scale, with higher scores representing a higher amount of the construct.
  Questions: How much do these messages...
  * make you concerned about the health effects of eating red meat?
  * make you concerned about the environmental effects of eating red meat?
  * discourage you from wanting to eat red meat?
  * make eating red meat seem unpleasant to you?
    1. Not at all, 2=Very little, 3=Somewhat, 4=Quite a bit, 5=A great deal).

SECONDARY OUTCOMES:
Attention | ~10 minute computer survey immediately after seeing messages
  How much the message grabs one's attention. Measured using a a 1 to 5 likert scale, with higher scores representing a higher amount of the construct.
Negative affect | ~10 minute computer survey immediately after seeing messages
  How much the messages make one feel scared. Measured using a a 1 to 5 likert scale, with higher scores representing a higher amount of the construct.
Cognitive elaboration | ~10 minute computer survey immediately after seeing messages
  How much the messages make one think about the environmental/health harms caused by eating meat. Measured using a a 1 to 5 likert scale, with higher scores representing a higher amount of the construct.
Social interactions | ~10 minute computer survey immediately after seeing messages
  How much one is likely to talk about the message with others in the next week. Measured using a 1 to 5 likert scale, with higher scores representing a higher amount of the construct.
Intention to reduce meat consumption | ~10 minute computer survey immediately after seeing messages
  How much one intends to reduce red meat consumption in the next 30 days. Measured using a a 1 to 5 likert scale, with higher scores representing a higher amount of the construct.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Rayala, Principal Investigator — University of North Carolina, Chapel Hill; Lindsey Smith Taillie, PhD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Population Center, Chapel Hill, North Carolina, United States

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT04562636/SAP_000.pdf